CLINICAL TRIAL: NCT00578669
Title: Sequential Use of Fluoxetine for Smokers With Elevated Depressive Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHI0710-002; 1R01DA023190 (NIH)
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Major Depressive Disorder; Nicotine Dependence; Depression
Keywords: Smoking Cessation; Tobacco Use Cessation; Antidepressants
MeSH Terms: conditions — Depressive Disorder, Major; Tobacco Use Disorder; Depression; Smoking Cessation; Tobacco Use Cessation | interventions — Fluoxetine; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Sequential antidepressant pharmacotherapy with (20mg) fluoxetine, begun 8 weeks prior to and extended throughout brief (behavioral) standard smoking cessation treatment with transdermal nicotine patch.
  Interventions: Drug: Fluoxetine
- 2 (Placebo Comparator): Sequential placebo medication (dextrose), begun 8 weeks prior to and extended throughout brief (behavioral) standard smoking cessation treatment with transdermal nicotine patch.
  Interventions: Drug: Dextrose

INTERVENTIONS:
Drug: Fluoxetine — 20mg once daily for 16 weeks
  Other Names: Prozac
  Arms: 1
Drug: Dextrose — Once daily for 16 weeks
  Arms: 2

SUMMARY:
The primary purpose of this study is to determine whether, among smokers with elevated depressive symptoms, sequential antidepressant pharmacotherapy with fluoxetine (20 mg) begun 8 weeks prior to and extended throughout standard smoking cessation treatment with transdermal nicotine patch (ST-TNP) will result in superior short-and long-term smoking cessation outcomes compared to sequential pharmacotherapy with placebo medication combined with ST-TNP. The secondary aim of the study is to test the hypothesis that, among smokers with elevated depressive symptoms, sequential treatment with fluoxetine will result in lower levels of depressive symptoms and negative mood and higher levels of positive mood immediately prior to and throughout the course of smoking cessation treatment relative to the placebo condition.

DETAILED DESCRIPTION:
Cigarette smoking is the leading cause of death and disability in the United States, accounting for over 430,000 deaths in this country every year. The selection hypothesis of smoking prevalence argues that smokers who are unable to quit successfully are likely to possess risk factors or characteristics that make it difficult to quit, such as nicotine dependence and psychiatric comorbidity. As such, significant strides in helping "today's" smokers quit will ultimately be found in the ability to develop specialized treatments that target the particular needs of subgroups of smokers, especially those who are at higher risk for relapse. Depression is the psychiatric disorder most frequently associated with cigarette smoking in adults and strong associations have been demonstrated between cigarette smoking and both depressive disorders and depressive symptoms. In fact, a prospective analysis from the National Health and Nutrition Examination Survey showed that smokers with elevated depressive symptoms were 40% less likely than nondepressed smokers to have quit nine years later.

The development of an efficacious, specialized treatment of nicotine dependence for smokers with elevated depressive symptoms would address this need by providing physicians with an effective treatment alternative for the large number of smokers with depressive symptoms seen daily in clinical practice. This study examines the hypothesis that smokers with elevated depressive symptoms treated with fluoxetine 8 weeks prior to quitting and extended throughout 8 weeks of standard treatment with the nicotine patch post-quit will demonstrate superior cessation outcomes compared to placebo medication combined with standard treatment and the nicotine patch, administered with the identical treatment schedule. A secondary hypothesis is to examine whether reductions in depressive symptoms and negative mood and increases in positive mood will be greater for those in the sequential fluoxetine versus placebo condition.

ELIGIBILITY:
Inclusion Criteria:

* Regular smoker for at least one year
* Currently smokes at least 10 cigarettes per day
* Elevated depressive symptoms
* Uses no other tobacco products

Exclusion Criteria:

* Current Axis I disorder, including Major Depressive Disorder
* Psychoactive substance abuse or dependence (excluding nicotine dependence) within past year
* Current use of psychotropic medication
* Use of antidepressant medication within past 6 months
* Current suicidal risk
* History of significant medical illness, such as cardiovascular disease, neurological, gastrointestinal, or other systemic illness
* Pregnancy or breast feeding
* Use of nicotine replacement therapy or of any medication for smoking cessation not provided by the researchers during the quit attempt

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2008-04; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Brown, Ph.D., Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website for Butler Hospital with links to research — http://www.butler.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequential Fluoxetine: Sequential Fluoxetine - Participants received sequential antidepressant pharmacotherapy (fluoxetine - 20 mg.) that was begun 8 weeks prior to, and extended throughout the treatment phase. The treatment phase consisted of 8 weeks of brief behavioral counseling and transdermal nicotine patches.
  Fluoxetine was used once daily for 16 weeks.
- Sequential Placebo: Sequential placebo medication (dextrose), begun 8 weeks prior to and extended throughout the 8-week brief (behavioral) standard smoking cessation treatment with transdermal nicotine patch.
  Dextrose was used once daily for 16 weeks
Period: Overall Study
Arm/Group | Sequential Fluoxetine | Sequential Placebo
Started | 107 | 99
Completed | 107 | 99
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequential Placebo: Participants received placebo medication, dextrose, that was begun 8 weeks prior to and extended throughout the brief, behavioral standard smoking cessation treatment that included transdermal nicotine patch.
  The placebo medication (dextrose) was taken once daily for 16 weeks.
- Sequential Fluoxetine: Participants received fluoxetine medication, 20 mg, that was begun 8 weeks prior to and extended throughout the brief, behavioral standard smoking cessation treatment that included transdermal nicotine patch.
  The fluoxetine medication (20 mg) was taken once daily for 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Sequential Placebo | Sequential Fluoxetine | Total
Number analyzed (Participants) | 99 | 107 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.05 (11.40) | 43.07 (10.97) | 43.54 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 51 | 99
  Male | 51 | 56 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 98 | 105 | 203
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 4
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 6 | 11
  White | 89 | 99 | 188
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 99 | 107 | 206
Cigarettes smoked per day (past month) [Mean (Standard Deviation); unit: cigarettes] | 21.07 (9.03) | 20.96 (10.33) | 21.01 (9.7)
Fagerstrom Test for Nicotine Dependence (FTND) [Mean (Standard Deviation); unit: units on a scale] — Scale can be scored on a range of 0 - 10. Higher scores signify greater levels of nicotine dependence.
  units on a scale | 5.40 (2.37) | 5.90 (1.74) | 5.66 (2.08)
Center for Epidemiologic Studies - Depression (CES-D) scale [Mean (Standard Deviation); unit: units on a scale] — CES-D consists of 20 items, with total scores on the scale ranging from 0 - 60. Higher scores are indicative of greater levels of depressive symptoms.
  units on a scale | 9.64 (8.53) | 9.90 (8.14) | 9.77 (8.31)
Center for Epidemiologic Studies - Depression (CES-D) > 16 [Count of Participants; unit: Participants] — CES-D consists of 20 items, with total scores on the scale ranging from 0 - 60. Higher scores are indicative of greater levels of depressive symptoms.
  Participants | 15 | 21 | 36
Recurrent major depressive disorder (MDD) [Count of Participants; unit: Participants] | 18 | 16 | 34
Single major depressive disorder (MDD) episode [Count of Participants; unit: Participants] | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Smoking Abstinence
Description: 7-day point prevalence abstinence
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Sequential Fluoxetine | Sequential Placebo
Number analyzed (Participants) | 107 | 99
Participants | 24 | 18

2. Secondary Outcome: Self-reported Depressive Symptoms
Description: Self-reported depressive symptoms based on the Center for Epidemiologic Studies-Depression (CES-D) scale. CES-D consists of 20 items, with total scores on the scale ranging from 0 - 60. Higher scores are indicative of greater levels of depressive symptoms.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sequential Fluoxetine | Sequential Placebo
Number analyzed (Participants) | 107 | 99
score on a scale | 9.9 (8.14) | 9.64 (8.53)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a one year period.
Description: Definitions of adverse event and/or serious adverse event do not differ from the clinicaltrials.gov definitions.
Groups:
- Sequential Fluoxetine: Sequential antidepressant pharmacotherapy with (20mg) fluoxetine, begun 8 weeks prior to and extended throughout brief (behavioral) standard smoking cessation treatment with transdermal nicotine patch.
  Fluoxetine: 20mg once daily for 16 weeks
- Sequential Placebo: Sequential placebo medication (dextrose), begun 8 weeks prior to and extended throughout brief (behavioral) standard smoking cessation treatment with transdermal nicotine patch.
  Dextrose: Once daily for 16 weeks
Arm/Group | Sequential Fluoxetine | Sequential Placebo
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/99
Other Adverse Events (participants affected / at risk) | 1/107 | 0/99
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sequential Fluoxetine (N=107) | Sequential Placebo (N=99)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No